CLINICAL TRIAL: NCT04250090
Title: Post-Marketing Follow-Up of Long-term Type Ureteral Stent Set
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: En Chu Kong Hospital (Other)
Responsible Party: Principal Investigator, ChungChengWang, Chief of urology, En Chu Kong Hospital
Other Study IDs: ECKIRB1050505
Record Dates: First submitted 2020-01-17; First posted 2020-01-31 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Ureter Stricture; Hydronephrosis
Keywords: Ureter Stricture; Hydronephrosis
MeSH Terms: conditions — Hydronephrosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Long-term type ureteral stent set: Patients with Long-term type ureteral stent set due to ureteral stricture.

SUMMARY:
Ureteral stents have been widely used in many urological operations. Although there are several reports regarding the effectiveness of long-term ureteral stents for malignancy ureteral obstruction, ureteral stricture and urolithiasis, the experience is limited about the long-term ureteral stents made by Taiwan. The investigators have to propose the 5-year post-market survey report. Though this observation study, The investigators can further understand the clinical safety and effectiveness of placing ureteral stents

DETAILED DESCRIPTION:
Ureteral stents have been widely used in many urological operations. The main purposes of placing ureteral stents include improvement of ureteral obstruction, protecting renal function and drainage of infection. Although there are several reports regarding the effectiveness of long-term ureteral stents for malignancy ureteral obstruction, ureteral stricture and urolithiasis, the experience is limited about the long-term ureteral stents made by Taiwan. Thus, The investigators will conduct this post-marketing survey to observe and investigate the changes of ureteral stents, e.g. hydronephrosis, infection and stone formation. Now this product has been approved by European Medical Device Administration. The investigators have to propose the 5-year post-market survey report. Though this observation study, The investigators can further understand the clinical safety and effectiveness of placing ureteral stents

ELIGIBILITY:
Inclusion Criteria:

1. Patients who used " Bioteq" Ureteral Stent Set (Long-Term Type) in their treatments.
2. Patients with complete basic parameters.

Exclusion Criteria:

1. Patients with any of the following conditions are excluded from this clinical study:

   Patients with incomplete basic parameters.
2. The minorities, children and special populations

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The most recent patients who actually used the " Bioteq" Ureteral Stent Set (Long-Term Type) are included, and a non-grouping method is adopted
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2019-07-09 (Actual); Primary Completion 2022-07-30 (Estimated); Study Completion 2022-10-31 (Estimated)

PRIMARY OUTCOMES:
Hydronephrosis | 5 years
  no hydronephrosis, mild hydronephrosis, moderate hydronephrosis, severe hydronephrosis
Renal function | 5 years
  serum BUN level
Renal function | 5 years
  serum Creatine level
Days of stent placement | 5 years
  Mean days of stent placement

CONTACTS AND LOCATIONS:
Overall Officials: Chung Cheng Wang, MD. Ph. D, Principal Investigator — Deputy Superintendent of Department of Education and Research
Locations (1):
- En Chu Kong Hospital, New Taipei City, Sanxia Dist., Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Liatsikos EN, Kagadis GC, Barbalias GA, Siablis D. Ureteral metal stents: a tale or a tool? J Endourol. 2005 Oct;19(8):934-9. doi: 10.1089/end.2005.19.934. PMID 16253054
- [Result] Zeljko M, Markovic B, Mladenovic A, Mijailovic M, Lukic S. Balloon dilatation and insertion of temporary coated stents using a retrograde approach in patients with irreversible strictures of the distal ureter. Jpn J Radiol. 2010 Nov;28(9):695-9. doi: 10.1007/s11604-010-0485-2. Epub 2010 Nov 27. PMID 21113756
- [Result] Bach T, Geavlete B, Herrmann TW, Gross AJ. Retrograde blind endoureterotomy for subtotal ureteral strictures: a new technique. J Endourol. 2008 Nov;22(11):2565-70. doi: 10.1089/end.2008.0173. PMID 19046096
- [Result] Aytekin C, Boyvat F, Harman A, Ozyer U, Colak T, Haberal M. Percutaneous therapy of ureteral obstructions and leak after renal transplantation: long-term results. Cardiovasc Intervent Radiol. 2007 Nov-Dec;30(6):1178-84. doi: 10.1007/s00270-007-9031-8. Epub 2007 May 17. PMID 17508243
- [Result] Kim BM, Park SI. Placement of double-J ureteric stent using the pull-through technique in patients with tight ureteric stenosis. Abdom Imaging. 2008 Mar-Apr;33(2):237-40. doi: 10.1007/s00261-007-9233-1. PMID 17440767
- [Result] Juaneda B, Alcaraz A, Bujons A, Guirado L, Diaz JM, Marti J, de la Torre P, Sabate S, Villavicencio H. Endourological management is better in early-onset ureteral stenosis in kidney transplantation. Transplant Proc. 2005 Nov;37(9):3825-7. doi: 10.1016/j.transproceed.2005.09.199. PMID 16386552
- [Result] Egilmez T, Guvel S, Kilinc F, Yaycioglu O, Ozkardes H. Management of complete ureteral obstructions with a transluminal puncture technique. Int Braz J Urol. 2005 May-Jun;31(3):264-8. doi: 10.1590/s1677-55382005000300013. PMID 15992432
- [Result] Uthappa MC, Cowan NC. Retrograde or antegrade double-pigtail stent placement for malignant ureteric obstruction? Clin Radiol. 2005 May;60(5):608-12. doi: 10.1016/j.crad.2004.11.014. PMID 15851050
- [Result] Unsal A, Cimentepe E, Balbay MD. Routine ureteral dilatation is not necessary for ureteroscopy. Int Urol Nephrol. 2004;36(4):503-6. doi: 10.1007/s11255-004-0860-y. PMID 15787325
- [Result] Mattei A, Danuser H. [Stents in urology]. Ther Umsch. 2003 Apr;60(4):233-7. doi: 10.1024/0040-5930.60.4.233. German. PMID 12731434
- [Result] Barbalias GA, Liatsikos EN, Kalogeropoulou C, Karnabatidis D, Zabakis P, Athanasopoulos A, Perimenis P, Siablis D. Externally coated ureteral metallic stents: an unfavorable clinical experience. Eur Urol. 2002 Sep;42(3):276-80. doi: 10.1016/s0302-2838(02)00281-6. PMID 12234513
- [Result] Hibi H, Kato K, Mitsui K, Taki T, Yamada Y, Honda N, Fukatsu H. Endoscopic ureteral incision using the holmium:YAG laser. Int J Urol. 2001 Dec;8(12):657-61. doi: 10.1046/j.1442-2042.2001.00393.x. PMID 11851764
- [Result] Micali S, De Carli P, Miano R, O'Sullivan D, Lamanna L, Micali F. Double-J ureteral stents: an alternative to external urinary stents in orthotopic bladder substitution. Eur Urol. 2001 May;39(5):575-9. doi: 10.1159/000052506. PMID 11464040
- [Result] Lin DW, Bush WH, Mayo ME. Endourological treatment of ureteroenteric strictures: efficacy of Acucise endoureterotomy. J Urol. 1999 Sep;162(3 Pt 1):696-8. doi: 10.1097/00005392-199909010-00017. PMID 10458345
- [Result] Puppo P, Ricciotti G, Bozzo W, Introini C. Primary endoscopic treatment of ureteric calculi. A review of 378 cases. Eur Urol. 1999;36(1):48-52. doi: 10.1159/000019926. PMID 10364655
- [Result] Ravery V, de la Taille A, Hoffmann P, Moulinier F, Hermieu JF, Delmas V, Boccon-Gibod L. Balloon catheter dilatation in the treatment of ureteral and ureteroenteric stricture. J Endourol. 1998 Aug;12(4):335-40. doi: 10.1089/end.1998.12.335. PMID 9726399
- [Result] Zimskind PD, Fetter TR, Wilkerson JL. Clinical use of long-term indwelling silicone rubber ureteral splints inserted cystoscopically. J Urol. 1967 May;97(5):840-4. doi: 10.1016/S0022-5347(17)63130-6. No abstract available. PMID 6025928
- [Result] Richter S, Ringel A, Shalev M, Nissenkorn I. The indwelling ureteric stent: a 'friendly' procedure with unfriendly high morbidity. BJU Int. 2000 Mar;85(4):408-11. doi: 10.1046/j.1464-410x.1998.00543.x-i1. PMID 10691815
- [Result] Pocock RD, Stower MJ, Ferro MA, Smith PJ, Gingell JC. Double J stents. A review of 100 patients. Br J Urol. 1986 Dec;58(6):629-33. doi: 10.1111/j.1464-410x.1986.tb05900.x. PMID 3801820
- [Result] Saltzman B. Ureteral stents. Indications, variations, and complications. Urol Clin North Am. 1988 Aug;15(3):481-91. PMID 3043868
- [Result] Ahallal Y, Khallouk A, El Fassi MJ, Farih MH. Risk factor analysis and management of ureteral double-j stent complications. Rev Urol. 2010 Spring;12(2-3):e147-51. PMID 20811552
- [Result] Lam JS, Gupta M. Tips and tricks for the management of retained ureteral stents. J Endourol. 2002 Dec;16(10):733-41. doi: 10.1089/08927790260472881. PMID 12542876
- [Result] Borboroglu PG, Kane CJ. Current management of severely encrusted ureteral stents with a large associated stone burden. J Urol. 2000 Sep;164(3 Pt 1):648-50. doi: 10.1097/00005392-200009010-00007. PMID 10953117
- [Result] Mohan-Pillai K, Keeley FX Jr, Moussa SA, Smith G, Tolley DA. Endourological management of severely encrusted ureteral stents. J Endourol. 1999 Jun;13(5):377-9. doi: 10.1089/end.1999.13.377. PMID 10446801
- [Result] Schulze KA, Wettlaufer JN, Oldani G. Encrustation and stone formation: complication of indwelling ureteral stents. Urology. 1985 Jun;25(6):616-9. doi: 10.1016/0090-4295(85)90293-6. PMID 4012953
- [Result] el-Faqih SR, Shamsuddin AB, Chakrabarti A, Atassi R, Kardar AH, Osman MK, Husain I. Polyurethane internal ureteral stents in treatment of stone patients: morbidity related to indwelling times. J Urol. 1991 Dec;146(6):1487-91. doi: 10.1016/s0022-5347(17)38146-6. PMID 1942324
- [Result] Somers WJ. Management of forgotten or retained indwelling ureteral stents. Urology. 1996 Mar;47(3):431-5. doi: 10.1016/S0090-4295(99)80468-3. PMID 8633417
- [Result] Singh I, Gupta NP, Hemal AK, Aron M, Seth A, Dogra PN. Severely encrusted polyurethane ureteral stents: management and analysis of potential risk factors. Urology. 2001 Oct;58(4):526-31. doi: 10.1016/s0090-4295(01)01317-6. PMID 11597531
- [Result] Kilciler M, Erdemir F, Bedir S, Coban H, Erten K, Guven O, Topac H. Spontaneous ureteral stent fragmentation: a case report and review of the literature. Kaohsiung J Med Sci. 2006 Jul;22(7):363-6. doi: 10.1016/S1607-551X(09)70324-9. PMID 16849106